CLINICAL TRIAL: NCT07068555
Title: Development of Prostate Cancer Dendritic Cell Vaccines
Brief Title: Prostate Cancer Vaccines
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-25002
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer Indications
Keywords: DC vaccine therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Immunomodulatory DC vaccines to target prostate cancer (Experimental): Prostate tumor antigen-modified autologous DCs
  Interventions: Biological: Immunomodulatory DC vaccines to target prostate cancer

INTERVENTIONS:
Biological: Immunomodulatory DC vaccines to target prostate cancer — 1 to 2 injections, with an interval of one month, of 1~2x10^7 DC vaccine administered subcutaneously

SUMMARY:
Tumor antigens are protein fragments produced by cancer cells carrying genetic mutations, and many tumor antigens are similar to normal protein antigens, making them unrecognizable by the immune system. Many tumor vaccines are prepared based on a single tumor antigen. This study is based on multiple target antigens using tumor lysates or synthetic peptides. The immune modulation by dendritic-cell (DC)-based cancer vaccines consists of genetically modified DCs to activate T cells to target cancer cells. The study is based on an advanced cancer vaccine technology, which aims to evaluate the safety and potential benefit of the novel immunomodulatory prostate cancer DC vaccines.

DETAILED DESCRIPTION:
Prostate cancer is a malignancy originating from the epithelial cells of the prostate gland, ranking as the second most common cancer among men worldwide. Its etiology involves factors such as genetics, age, lifestyle (e.g., high-fat diet, obesity), and hormone levels. High-risk populations are typically men aged 45 and above.

Prostate cancer vaccines based on multiple target antigens derived from tumor lysates or synthetic peptides can serve as antigenic targets for immune cells. The vaccines involve immunomodulation with autologous DCs to stimulate and activate T cells in the body to target cancer cells. The principle of the DC vaccines is simple: to harness and enhance the body's anti-cancer immunity. The process involves simulating antigen-presenting cells with target tumor antigens in culture and then injecting patients with the modified antigen-presenting DCs. Early studies of DC-based vaccines targeting prostate cancer have shown high safety and low toxicity. Here, the study aims to evaluate the safety and efficacy of prostate cancer DC vaccines that use multiple target antigens based on prostate cancer cells to stimulate and induce a specific and strong anti-cancer immune response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* WBC ≥ 3,500/µL
* Platelet count ≥ 100,000/µL
* Hemoglobin ≥ 10.0 g/dL
* Creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 2.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Fertile patients must use effective contraception
* Willing to provide blood samples for research purposes
* Able to complete questionnaire(s) alone or with assistance
* Able to undergo leukapheresis
* No known immunodeficiency
* No other malignancy within the past 5 years except for basal cell or squamous cell carcinoma of the skin treated with local resection only
* No concurrent serious illness
* No known history of positive PPD skin test
* Human immunodeficiency virus (HIV) and Hepatitis C virus (HCV) test negative.

Exclusion Criteria:

* The patient was still using dexamethasone at a dose greater than 4 mg/day during mononuclear cell collection
* Patients have a history of autoimmune diseases or other diseases requiring long-term use of hormones or immunosuppressive drugs
* Patients with a history of allergies or allergies to immune cells and adjuvants of cellular products
* Active infection with fever
* Patients with neutropenia (> 10 days) that are difficult to correct after treatment
* Infection with bacteria, fungi or viruses, uncontrolled
* Patients with HIV and those living with active HBV and HCV
* Severe organ failure (heart, liver, kidney, lung)
* Patients who had previously been treated with cell therapy products and examined by team experts deemed not suitable for treatment
* Anything that researchers believe may increase the risk of subjects or interfere with test results

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Events of adverse effects after the DC vaccine injection | up to one month
  To assess the safety of autologous prostate cancer DC vaccine in vivo. The percentage of patients who have adverse effects will be evaluated by using the NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Rate of successful prostate cancer DC vaccine generation | up to one month
  The percentage of successful prostate cancer DC vaccine generation, which are derived from the monocytic cells of the subjects and pass the safety test after standard culture procedures, viable for at least one preparation, will be evaluated.
Ability of prostate cancer DC vaccines to induce anti-cancer reaction | after 1 month from prostate cancer DC injection to 12 months after injection
  Measurement of specific T cell concentration in blood sample
Ability of prostate cancer DC vaccines to induce an anti-cancer reaction | after 1 month from prostate cancer DC injection to 24 months after injection
  Objective response complete response (CR) is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. CR indicates disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have shown reduction in short axis to <10 mm.
Ability of prostate cancer DC vaccines to induce an anti-cancer reaction | after 1 month from prostate cancer DC injection to 24 months after injection
  Objective response partial response (PR)) is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No